CLINICAL TRIAL: NCT06441084
Title: A Phase I or II Clinical Trial Evaluating the Safety and Efficacy of NCR300 Injection in Preventing Recurrence of Acute Myeloid Leukemia After Allogeneic Blood Stem Cell Transplantation
Brief Title: A Trial to Evaluate the Safety and Efficacy of NCR300 in Preventing Recurrence of Acute Myeloid Leukemia（AML) After Transplantation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCR300-2002
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: iNK
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCR300 injection (Experimental): Cohort1: Low dose NCR300 injection; Cohort2: Mid-low dose NCR300 injection; Cohort3: Mid-high dose NCR300 injection; Cohort4: High dose NCR300 injection.
  Interventions: Biological: NCR300 injection

INTERVENTIONS:
Biological: NCR300 injection — Subjects will receive at least 1 cycle of NCR300 injection.

SUMMARY:
A Trial to Evaluate the Safety and Efficacy of iNK in the Treatment of Subjects for Preventing Recurrence of Acute Myeloid Leukemia After Allogeneic Blood Stem Cell Transplantation.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability and preliminary efficacy of NCR300 injection.

ELIGIBILITY:
Inclusion Criteria:

1.Subjects who understand and voluntarily sign the Informed Consent Form(ICF);

2.18-65years;

3.Clinical diagnosis of AML;

4.Accepted allogeneic blood stem cell transplantation within 60 to 28 days prior before initial infusion;

5.Complete donor chimerism and with high-risk recurrence factors prior to transplantation , or bone marrow examination shows positive MRD；

6.Have already recovered from the adverse reactions of previous treatment；

7.Having appropriate organ functions；

8.Eastern Cooperative Oncology Group(ECOG)<3;

9.Subjects who are able to comply with contraceptives from the study period to 6 months after the end of this study;

Exclusion Criteria:

1. Bone marrow examination shows hematological recurrence;
2. Have malignant tumors within 5 years before screening;
3. Subjects with acute promyelocytic leukemia(APL);
4. Subjects with severe respiratory diseases;
5. Subjects with clear history of neurological or psychiatric disorders in the past;
6. Active central nervous system involvement；
7. HIV(human immunodeficiency virus) antibody positive,treponema pallidum(TP) antibody positive.Have active hepatitis B or hepatitis C;
8. Allergies to NCR300 or its excipients;
9. Subjects with active cardiovascular and cerebrovascular diseases;
10. Received organ transplantation or planned transplantation；
11. Received other treatment drugs after transplantation；
12. Graft-Versus-Host Disease (GVHD)>II grades;
13. Subjects with active nervous system autoimmune or inflammatory diseases;
14. Expected survival period within 3 months;
15. Have alcohol or drug addiction or with a clear history of mental disorders or with a history of drug abuse or drug use of psychotropic substances;
16. Having mental illness；
17. Having uncontrollable active infections;
18. Subjects whose state is not suitable for entering the study;
19. Other situations determined by investigator that it is not suitable to enter the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity(DLT) | 4 weeks after initial infusion
  Number of participants with Dose-limiting toxicity in 28 days after first infusion
Adverse Event(AE) or Serious Adverse Event(SAE) | From the date of initial infusion to a year after initial infusion
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Maximum plasma concentration(Cmax) | 2 hours before initial infusion;4 hours ,24 hous, 3 Days after initial infusion.2 hours before second infusion; 24 hous, 3 Days after second infusion.
  Maximum plasma concentration of NCR300 in peripheral blood
Time after doing at which maximun plasma concentration is reached(Tmax) | 2 hours before initial infusion;4 hours ,24 hous, 3 Days after initial infusion.2 hours before second infusion; 24 hous, 3 Days after second infusion.
  Time after doing at which maximun plasma concentration of NCR300 in peripheral blood is reached
Cumulative Incidence of Relapse(CIR) | 6 Months After Initial Infusion
  The proportion of patients with hematological recurrence within 6 months after initial infusion to all patients
Minimal Residual Disease(MRD) | From the date of screening to a year after initial infusion
  Changes in MRD before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Doctor, Principal Investigator — Capital Medical University